CLINICAL TRIAL: NCT04029363
Title: Expanded Study of the HighLife 28mm Trans-septal Trans-catheter Mitral Valve in Patients With Moderate-severe or Severe Mitral Regurgitation and at High Surgical Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HighLife SAS (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-2018-01-TS Expanded EU/AU
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): Single arm, non-randomized
  Interventions: Device: HighLife Transcatheter Mitral Valve Replacement

INTERVENTIONS:
Device: HighLife Transcatheter Mitral Valve Replacement — Transcatheter Mitral Valve Replacement

SUMMARY:
to evaluate the safety and performance of the HighLife 28mm transcatheter, trans-septal Mitral Valve in patients with moderate-severe or severe mitral regurgitation who are at high risk for surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years 2. Moderate-severe or severe mitral regurgitation (≥ 3+) 3. Patient has New York Heart Association (NYHA) Functional Class II, III or ambulatory IV 4. Patient is under guideline directed medical therapy, as reviewed and confirmed by the local multidisciplinary Heart Team, for at least one month 5. Patient is high-risk for open-heart surgery based on the assessment of the multidisciplinary Heart Team using standard scoring systems and consideration of co-morbidities, frailty, and disability 6. Patient meets the anatomical criteria for HighLife valve 7. Patient is willing to participate in the study and provides signed informed consent

Exclusion Criteria:

1. Any stroke/TIA within 30 days
2. Severe symptomatic carotid stenosis (> 70% by non-invasive imaging)
3. Active infections requiring antibiotic therapy
4. Active ulcer or gastro-intestinal bleeding in the past 3 months
5. History of bleeding diathesis, coagulopathy or refusal of future blood transfusion
6. Patients in whom TEE is not feasible
7. Patients who are pregnant or lactating, or plan to get pregnant in the next 12 months.
8. Patient is unable to comply with the follow-up schedule and assessments
9. Participation in another clinical investigation at the time of inclusion
10. Patient has known allergies to the device components or contrast medium
11. Patient cannot tolerate anticoagulation or antiplatelet therapy
12. Patients with a life expectancy of less than 12 months due to non-cardiac conditions
13. Patient had permanent pacemaker, or similar device with implantable cardiac leads (i.e. resynchronization therapy) within the last 3 months

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2031-12-15 (Estimated)

PRIMARY OUTCOMES:
Device Safety | 30 days
  Freedom from major adverse events

CONTACTS AND LOCATIONS:
Locations (50):
- Australia (11):
  - St. Vincent's Hospital - Sydney, Darlinghurst, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - St. Andrew's Hospital, Adelaide
  - Princess Alexandra Hospital, Brisbane
  - Warringal Hospital, Heidelberg
  - The Alfred Hospital, Melbourne
  - John Hunter Hospital, Newcastle
  - Mount Hospital, Perth
  - North Shore Private Hospital, Sydney
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan, Bruges
  - UZ Leuven, Leuven
- France (12):
  - Rangueil University Hospital, Toulouse, Toulouse
  - CHU Lille, Lille
  - Medipole Lyon-Villeurbanne, Lyon
  - Hopital Prive - Jacques Cartier, Massy
  - Centre Hospitalo-Universitaire de Nantes, Nantes
  - European Hospital George Pompidou, Paris
  - CHU Bordeaux, Pessac
  - CHU de Rennes, Rennes
  - Centr Cardiologiqque du Nord, Saint-Denis
  - CHRU Strasbourg, Strasbourg
  - Clinque Pasteur, Toulouse
  - Rangueil University Hospital, Toulouse
- Germany (10):
  - University Heart Center Freiburg - Bad Krozingen, Bad Krozingen
  - Universitaetsklinikum Bonn, Bonn
  - Heart Center, University Hospital Dresden, Dresden
  - Universitatsklink Hamburg-Eppendorf, Hamburg
  - Mediinisches Versorgungszentrum, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Herzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum Munchen, Munich
  - University Medicine Dept of Cardiology, Rostock
  - University Hospital Ulm, Ulm
- Poland (5):
  - Medical University of Gdansk, Gdansk
  - Medical University of Silesia Hospital, Katowice
  - University Hospital of Lord's Transfiguration, Poznan
  - Medical University of Warsaw, Warsaw
  - Institute of Cardiology, Warsaw
- National Heart Center Singapore, Singapore, Singapore
- United Kingdom (8):
  - Royal Victoria Hospital, Belfast
  - Brighton and Sussex University Hospital, Brighton
  - Royal Infirmary of Edinburgh, Edinburgh
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Guy's and St. Thomas' NHS Foundation Trust - St. Thomas Hospital, London
  - Barts Heart Center, London
  - John Radcliffe, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider LM, Worthley S, Nickenig G, Huczek Z, Wojakowski W, Tchetche D, Dubois C, Nasr M, Verhees L, Rothman M, Piazza N, Buithieu J, Yeow WL, Kessler M, Rottbauer W. 1-Year Outcomes Following Transfemoral Transseptal Transcatheter Mitral Valve Replacement: The HighLife TSMVR Feasibility Study. JACC Cardiovasc Interv. 2023 Dec 11;16(23):2854-2865. doi: 10.1016/j.jcin.2023.09.003. Epub 2023 Nov 22. PMID 37999708